CLINICAL TRIAL: NCT05198635
Title: Association Between Local Cerebral Oxygen Saturation Monitoring and Postoperative Delirium in Carotid Endarterectomy：A Prospective Cohort Study
Brief Title: Association Between Local Cerebral Oxygenation Monitoring and Postoperative Delirium in Carotid Endarterectomy
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Prof., Beijing Tiantan Hospital
Other Study IDs: 20220105
Record Dates: First submitted 2022-01-04; First posted 2022-01-20 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Oxygen Saturation; Postoperative Delirium; Carotid Endarterectomy
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Device: local cerebral oxygen saturation
- Group 2
  Interventions: Device: local cerebral oxygen saturation

INTERVENTIONS:
Device: local cerebral oxygen saturation — minimum SctO2, SctO2 drop/rise defined by different thresholds, and area under/above the threshold

SUMMARY:
Postoperative delirium (POD) is a common perioperative complication, which can lead to adverse outcomes. Patients undergoing carotid endarterectomy (CEA) were elderly, complicated with vascular risk factors, cognitive dysfunction, some also had a history of stroke, and the circulation fluctuated greatly during the operation, often resulting in hypoperfusion of cerebral tissue and hypoxia. Therefore, they're the high-risk group of POD. Near-infrared Spectroscopy (NIRS) can continuously and noninvasively monitor local cerebral oxygen saturation (SctO2) to identify the mismatch of oxygen supply and demand in brain tissue. However, for CEA patients, the association between intraoperative SctO2 changes and POD remains unclear. This study intends to explore the association between them and determine the SctO2 threshold for predicting POD. We will monitor SctO2 intraoperatively, follow up and collect data postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Scheduled carotid endarterectomy; Signed informed consent.

Exclusion Criteria:

Severe cognitive impairment(Mini-Mental State Examination, MMSE<18); History of psychotropic drugs; Previous intracranial surgery history; Poor hearing or vision; Language barriers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Scheduled carotid endarterectomy
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | With postoperative 5 day
  Postoperative delirium is assessed by the Confusion assessment method for intensive care unit (CAM-ICU) or the 3-minute diagnostic interview for CAM (3D-CAM) when the patient is in intensive care unit or general ward, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Yuming MD Peng, Ph.D, Principal Investigator — Beijing Tian Tan Hospital
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No